CLINICAL TRIAL: NCT04984213
Title: CORTI-FIX: Clinical and Radiographic Outcomes Following Lumbar Interbody Placement With Posterior Minimally Invasive Intra-Laminar PEEK Ratcheting Fixation Device
Brief Title: Study of the Long-Term Outcomes of Posterior Spinal Fixation With the Karma Device
Status: Completed | Type: Observational
Sponsor: Spinal Elements (Industry)
Responsible Party: Sponsor
Other Study IDs: SEI-004
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Disc Disease
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Karma Posterior Fixation Device — Posterior Fixation

SUMMARY:
The primary objective of this clinical study is to measure fusion rate in patients at 12 months following lumbar fusion in combination with posterior fixation using the Karma® device.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature and age ≥ 18 years of age
2. Appropriate patient as determined by the Investigator for anterior or lateral approach to lumbar interbody fusion surgery with planned posterior fixation to treat degenerative disc disease in one or two adjacent vertebral levels between L2 and S1.
3. Failed at least six months of conservative treatment. This may or may not include any of the following,

   1. Spinal injections
   2. Chiropractic care
   3. Physical therapy
   4. Activity modification and/or with anti-inflammatory medications
4. Oswestry Low Back Pain Disability Questionnaire score of at least 30%
5. Visual Analog Scale (VAS) for back/hip/lower extremity pain ranking at a minimum at least 3/10 (30%)
6. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule, study requirements with a signed informed consent with a study collaborator present at the time of signing to ensure compliance.

Exclusion Criteria:

1. Patients with greater than two levels of degenerative disease or deformity for INTENDED operative levels.
2. Previous fusion or total disc replacement at the intended level/s
3. Known allergy to implant and instrument materials
4. Clinically compromised vertebral bodies at the affected level(s) due to current or past trauma
5. Degenerative spondylolisthesis of grade >2
6. Isthmic spondylolisthesis
7. Back or leg pain of unknown etiology
8. Active systemic infection or infection at the location planned surgery
9. Active or suspected malignancy. If symptom free for 2 years, patients with prior malignancy may be included.
10. Morbid obesity defined as a body mass index > 40
11. Patient being treated for other specific medical conditions that may affect bone density or the ability to obtain fusion (ie: steroids, etc)
12. Pregnant or have plans to become pregnant in the next year.
13. Currently a prisoner
14. Patient has any condition, that in the opinion of the Investigator, would prohibit the patient from complying with the protocol
15. Participation in a concurrent clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects needing a lumbar fusion surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Fusion Rate | 12 months
  Interbody Fusion Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Spine Institute of Louisiana, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No